CLINICAL TRIAL: NCT07118072
Title: Internet-Delivered Skills Training in Affective and Interpersonal Regulation (i-STAIR) for Individuals With Adverse Childhood Experiences and Subsyndromal Depression: A Pilot Study
Brief Title: A Pilot Study to Examine the Efficacy of Internet-Delivered Skills Training in Affective and Interpersonal Regulation (i-STAIR) for Individuals With Adverse Childhood Experiences and Subsyndromal Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-3342
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Subthreshold Depression
Keywords: skills training in affective and interpersonal regulation; emotion regulation; subthreshold depression; prevention intervention; digital intervention; transdiagnostic intervention; Singapore
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized into two groups: Active intervention (i-STAIR; n = 75) or control (online general psychoeducation; n =75) groups. The active intervention group will receive a free 8-week (i.e., eight online sessions; 1 session per week) i-STAIR intervention and the control group will receive online psychoeducation intervention (i.e., 5 online sessions and three self-guided activities over 8 weeks). All interventions will be delivered online over Zoom or Microsoft Teams. All participants will complete the assessment measures (i.e., emotion dysregulation, interpersonal skills, perceptions of social support, depressive symptoms, and PTSD symptoms) at baseline, mid-intervention (i.e., four weeks), post-intervention (i.e., eight weeks).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Delivered Skills Training in Affective and Interpersonal Regulation (Experimental): i-STAIR specifically targets emotion dysregulation and poor interpersonal skills. i-STAIR comprises eight sessions (one hour per session, per week) and each session focuses on a particular skills deficit. In general, session-by-session topics include: (1) labelling and identifying feelings; (2) emotion management (i.e., focus on anger and anxiety); (3) distress tolerance; (4) acceptance of feelings and enhanced experiencing of positive emotions; (5) identification of trauma-based interpersonal schemas and their enactment in day-to-day life; (6) identification of conflict between trauma-generated feelings and current interpersonal goals; (7) role plays related to issues of power and control; and (8) role plays related to developing flexibility in interpersonal situations involving power differentials.
  Interventions: Behavioral: Internet-Delivered Skills Training in Affective and Interpersonal Regulation
- Online general psychoeducation (Active Comparator): Online general psychoeducation comprises five online sessions (one hour per session on Week 1, Week 2, Week 4, Week 6, and Week 8) where a trained research staff will provide psychoeducation to the participant for up to 1 hour, as well as three weeks of self-guided activities where the participant will work on a specific activity on their own and feedback will be provided during the online sessions. The online psychoeducation content will focus on the link between adverse childhood experiences and depression, and healthy lifestyle changes including healthy diet, exercise, and sleep.
  Interventions: Behavioral: Online general psychoeducation

INTERVENTIONS:
Behavioral: Internet-Delivered Skills Training in Affective and Interpersonal Regulation — Internet-Delivered Skills Training in Affective and Interpersonal Regulation (i-STAIR) is a psychological intervention that is focused on applying skills to improve emotion regulation difficulties and reduce interpersonal problems over two months (eight sessions; one session per week). i-STAIR also significantly reduces PTSD symptoms without direct discussion of the trauma and may be used alone or adjunctively to boost the effects of trauma-focused therapies.
  Arms: Internet-Delivered Skills Training in Affective and Interpersonal Regulation
Behavioral: Online general psychoeducation — Online general psychoeducation will focus on the teaching the link between adverse childhood experiences and depression, as well as teaching healthy lifestyle changes involving diet, exercise, and sleep. The online general psychoeducation will involve engaging presentations, active discussions, and self-directed homework activities.
  Arms: Online general psychoeducation

SUMMARY:
The present study aims to pilot internet-delivered Skills Training in Affective and Interpersonal Regulation (i-STAIR) as a transdiagnostic emotion dysregulation intervention to prevent progression to depression in individuals with adverse childhood experiences (ACEs) and subsyndromal depression. The aims of the study are: (i) to examine the effectiveness of i-STAIR on emotion dysregulation, interpersonal skills, depressive and PTSD symptoms at post-intervention i.e. on completion of the intervention (8 weeks); (ii) to examine if gains were maintained at 3 month post- intervention follow-up.

DETAILED DESCRIPTION:
Internet-delivered Skills Training in Affective and Interpersonal Regulation (i-STAIR) will be an effective intervention for preventing depression among those with adverse childhood experiences and subsyndromal depression. In contrast to the control group (i.e., individuals who received online general psychoeducation), we hypothesize that participants who receive i-STAIR will experience a significant reduction of depressive/PTSD symptoms and emotion dysregulation, as well as experience significant positive increases in interpersonal skills and perceptions of social support at post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to mild, moderate or severe adverse childhood experiences (ACEs)
* Screened positive for subsyndromal depression
* Singapore citizens or permanent residents (PRs)
* Aged 21 years to 65 years
* Able to speak and understand English
* Willing and able to undergo intervention and assessment online

Exclusion Criteria:

* Currently diagnosed with any mental disorder diagnoses;
* Experience cognitive impairment as determined by attending physician
* Have received or currently receiving dialectical behavior therapy (DBT) due to similarities with i-STAIR
* Female participants who are pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The Patient Health Questionnaire 9 | From enrollment to the end of follow-up at 20 weeks.
  The PHQ-9 will be used to assess for self-reported depressive symptoms. The PHQ-9 comprises 9 items which are rated on a 4-point Likert scale (ranging from 0=not at all to 3=nearly every day). Higher scores indicate more severe depressive symptoms. The PHQ-9 is used in the local clinical setting for routine screening of depressive symptoms.
Difficulties with Emotion Regulation Scale Short | From enrollment to the end of follow-up at 20 weeks.
  The DERS-S will be used to assess for global emotion dysregulation. Global emotion dysregulation comprises 6 dimensions: non-acceptance of emotional response, difficulties engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. Higher scores will indicate more severe global emotion dysregulation.
Ruminative Response Scale short-form | From baseline to end of follow-up at 20 weeks.
  The RRS will be used to measure habitual rumination. Rumination is a prevalent maladaptive emotion regulation strategy among patients with mental disorders and exerts a moderate to strong effect on psychopathology. Higher scores on the RRS will indicate more frequent use of rumination. The RRS demonstrated good psychometric properties in the literature.
Multidimensional Scale of Perceived Social Support | From baseline to end of follow-up at 20 weeks.
  The MSPSS will be used to measure an individual's level of perceived social support from three sources: Significant Others, Family and Friends. The MSPSS comprises 12 items and each item is rated on a seven-point Likert-type scale (ranging from 1=Very Strongly Disagree to 7=Very Strongly Agree).
Positive Mental Health Instrument | From baseline to end of follow-up at 20 weeks.
  The PMHI will be used to measure interpersonal skills. The PMHI and its subscales have been locally validated and demonstrated good psychometric properties in previous studies.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 | From baseline to end of follow-up at 20 weeks.
  The PCL-5 will be used to assess for self-reported PTSD symptoms. The PCL-5 is self-rated and higher scores indicate more severe PTSD symptoms (total score range from 0 to 80).
Work Productivity and Activity Impairment Questionnaire Specific Health Problem V2.0 | At baseline and post-intervention at 8 weeks only.
  The WPAI will be used to assess for the impact of health problems (e.g. physical or mental) on an individual's ability to work and perform regular activities. The WPAI: SHP comprises 1 dichotomous (yes/no) item asking if the respondent is currently employed, 3 items asking about the number of hours that the respondent worked or did not work in the past week, and 2 eleven-point Likert-type scales (ranging from 0 to 10; higher scores indicate more problems) asking about how much health problems affected the respondent's work productivity and ability to do regular daily activities.
Session Rating Scale | At mid-intervention at 4 weeks and at post-intervention at 8 weeks only.
  The SRS will be used to assess for therapeutic alliance between the participant and research therapist. The SRS has three scales that assess for the relational bond between participant and research therapist, goal agreement, and task agreement. An overall scale also assesses whether the participant felt that "there was something missing in the session" versus "overall the session was good for me". Overall, the SRS has a total of four scales and they are all assessed along a 100mm. Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mythily Subramaniam, MBBS, Ph.D., Study Director — Institute of Mental Health, Singapore; Siow Ann Chong, MD, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
The IPD will be subjected to review and ethical clearance by our ethics board. Hence, we may not be allowed to share IPD due to ethical requirements.

REFERENCES:
- [Background] Miu AC, Szentagotai-Tatar A, Balazsi R, Nechita D, Bunea I, Pollak SD. Emotion regulation as mediator between childhood adversity and psychopathology: A meta-analysis. Clin Psychol Rev. 2022 Apr;93:102141. doi: 10.1016/j.cpr.2022.102141. Epub 2022 Feb 21. PMID 35219929
- [Background] Subramaniam M, Abdin E, Seow E, Vaingankar JA, Shafie S, Shahwan S, Lim M, Fung D, James L, Verma S, Chong SA. Prevalence, socio-demographic correlates and associations of adverse childhood experiences with mental illnesses: Results from the Singapore Mental Health Study. Child Abuse Negl. 2020 May;103:104447. doi: 10.1016/j.chiabu.2020.104447. Epub 2020 Mar 12. PMID 32171798
- [Background] Hassija, C.M., and Cloitre, M. (2015). STAIR narrative therapy: a skills focused approach to trauma-related distress. Current Psychiatry Reviews, 11, 172-179.
- [Background] Karsten J, Penninx BW, Verboom CE, Nolen WA, Hartman CA. Course and risk factors of functional impairment in subthreshold depression and anxiety. Depress Anxiety. 2013 Apr;30(4):386-94. doi: 10.1002/da.22021. Epub 2012 Nov 16. PMID 23165799
- [Background] Kirlic N, Cohen ZP, Singh MK. Is There an Ace Up Our Sleeve? A Review of Interventions and Strategies for Addressing Behavioral and Neurobiological Effects of Adverse Childhood Experiences in Youth. Advers Resil Sci. 2020 Mar;1(1):5-28. doi: 10.1007/s42844-020-00001-x. Epub 2020 Mar 13. PMID 34278327
- [Background] Korotana LM, Dobson KS, Pusch D, Josephson T. A review of primary care interventions to improve health outcomes in adult survivors of adverse childhood experiences. Clin Psychol Rev. 2016 Jun;46:59-90. doi: 10.1016/j.cpr.2016.04.007. Epub 2016 Apr 21. PMID 27179348
- [Background] Liu J, Tan BCW, Abdin E, Padmini YS, Oh JY, Chong SA, Subramaniam M. Health care utilization, productivity losses, and burden of adverse childhood experiences in Singapore: Findings from a national survey. Psychol Trauma. 2025 Jan;17(1):1-9. doi: 10.1037/tra0001691. Epub 2024 Jun 20. PMID 38900512
- [Background] Lorenc T, Lester S, Sutcliffe K, Stansfield C, Thomas J. Interventions to support people exposed to adverse childhood experiences: systematic review of systematic reviews. BMC Public Health. 2020 May 12;20(1):657. doi: 10.1186/s12889-020-08789-0. PMID 32397975
- [Background] Cuijpers P, Pineda BS, Ng MY, Weisz JR, Munoz RF, Gentili C, Quero S, Karyotaki E. A Meta-analytic Review: Psychological Treatment of Subthreshold Depression in Children and Adolescents. J Am Acad Child Adolesc Psychiatry. 2021 Sep;60(9):1072-1084. doi: 10.1016/j.jaac.2020.11.024. Epub 2021 Feb 14. PMID 33596437
- [Background] Cloitre M, Koenen KC, Cohen LR, Han H. Skills training in affective and interpersonal regulation followed by exposure: a phase-based treatment for PTSD related to childhood abuse. J Consult Clin Psychol. 2002 Oct;70(5):1067-74. doi: 10.1037//0022-006x.70.5.1067. PMID 12362957
- [Background] Cloitre M, Garvert DW, Weiss BJ. Depression as a moderator of STAIR Narrative Therapy for women with post-traumatic stress disorder related to childhood abuse. Eur J Psychotraumatol. 2017 Oct 10;8(1):1377028. doi: 10.1080/20008198.2017.1377028. eCollection 2017. PMID 29038682
- See also: Related Info — https://www.predict-imhresearch.sg/